CLINICAL TRIAL: NCT00004132
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Recombinant Human Keratinocyte Growth Factor (rHuKGF) in Patients With Hematologic Malignancies Undergoing Total Body Irradiation (TBI) and High-Dose Chemotherapy With Autologous Peripheral Blood Progenitor Cell (PBPC) Transplantation
Brief Title: Growth Factor to Prevent Oral Mucositis in Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: AMGEN-KGF-980231-03; UCLA-9812041; CDR0000067362 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1609
Record Dates: First submitted 1999-12-10; First posted 2004-05-20 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Oral Complications; Radiation Toxicity
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; childhood Burkitt lymphoma; refractory multiple myeloma; stage 0 chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage IV childhood lymphoblastic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; oral complications; stage IV childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; primary central nervous system non-Hodgkin lymphoma; drug/agent toxicity by tissue/organ; radiation toxicity; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; anaplastic large cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Radiation Injuries; Hodgkin Disease; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Fibroblast Growth Factor 7; Cyclophosphamide; Etoposide; Ifosfamide; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: palifermin
Drug: cyclophosphamide
Drug: etoposide
Drug: ifosfamide
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Keratinocyte growth factor may prevent symptoms of mucositis in patients receiving radiation therapy and chemotherapy.

PURPOSE: Randomized phase II trial to study the effectiveness of keratinocyte growth factor in preventing oral mucositis in patients who have hematologic cancers and who are undergoing radiation therapy and chemotherapy before autologous peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of recombinant keratinocyte growth factor in reducing the duration of severe oral mucositis induced by total body irradiation and high dose chemotherapy in patients with hematologic malignancies. II. Determine the incidence and duration of severe oral mucositis, grade 2-4 diarrhea, and febrile neutropenia in these patients. III. Determine the necessity of use of transdermal or parenteral opioid analgesics and IV antifungals or antibiotics for febrile neutropenia or infections in these patients. IV. Determine the quality of life of these patients.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified by center. Patients are randomized to one of three treatment arms. Arm I: Patients receive 7 doses of recombinant human keratinocyte growth factor (rHuKGF). Arm II: Patients receive 4 doses of rHuKGF followed by 3 doses of placebo. Arm III: Patients receive 7 doses of placebo. Patients receive one of two conditioning regimens. Primary conditioning regimen: Patients receive rHuKGF or placebo daily on days -11, -10, -9, -5, 0, 1, and 2. Total body irradiation (TBI) is administered twice a day on days -8 to -5. Patients receive etoposide on day -4, cyclophosphamide IV over 1 hour on day -2, and peripheral blood stem cell transplantation (PBSCT) on day 0. Filgrastim (G-CSF) IV or SC is administered beginning on day 0 and continuing for 21 days or until blood counts recover. Secondary conditioning regimen: Patients receive rHuKGF or placebo daily on days -13, -12, -11, -7, 0, 1, and 2. TBI is administered twice a day on days -10 to -7. Patients receive ifosfamide IV over 1 hour followed by etoposide over 23 hours on days -6 to -2, then PBSCT on day 0. G-CSF IV or SC is administered beginning on day 0 for 21 days or until blood counts recover. Quality of life is assessed daily beginning on day -11 and continuing until day 28. Patients are followed at day 28 and then at day 60-100.

PROJECTED ACCRUAL: A minimum of 111 patients (37 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of Non-Hodgkin's lymphoma, Hodgkin's disease, acute myelogenous leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, chronic lymphocytic leukemia, or multiple myeloma Eligible for total body irradiation plus high dose chemotherapy followed by autologous peripheral blood stem cell transplantation At least 1,500,000 CD34+ cells/kg cryopreserved No prior treatment on this study

PATIENT CHARACTERISTICS: Age: 12 to 65 Performance status: Karnofsky 70-100% SWOG 0 or 1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1000/mm3 Platelet count greater than 100,000/mm3 If conditioning regimen scheduled soon after apheresis, platelet count of greater than 50,000/mm3 but less than 100,000/mm3 allowed Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No congestive heart failure No New York Heart Association class III or IV heart disease Pulmonary: DLCO at least 50% predicted Other: No prior or concurrent second malignancy No active infection or oral mucositis No insulin dependent diabetes mellitus HIV negative No sensitivity to E. coli derived products Not pregnant or nursing Fertile patients must use effective contraception one month before, during, and one month after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow or peripheral blood stem cell transplantation, unless undergoing second transplant of a tandem transplant regimen, with no complications after first transplant No concurrent interleukin-11 Chemotherapy: No other concurrent cytotoxic chemotherapy, except intrathecal methotrexate for CNS involvement Endocrine therapy: Not specified Radiotherapy: No prior extensive radiotherapy that would preclude total body irradiation Surgery: Not specified Other: At least 30 days since prior investigational devices or drugs, except Baxter Isolex i column No other concurrent investigational agents No concurrent prophylactic oral cryotherapy during chemotherapy

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States